CLINICAL TRIAL: NCT00583830
Title: A Phase 2, Randomized, Multi-Center, Open-Label Study to Evaluate the Efficacy and Safety of Mapatumumab in Combination With Carboplatin and Paclitaxel as First Line Therapy in Subjects With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Mapatumumab in Combination With Paclitaxel and Carboplatin in Subjects With Non-small Cell Lung Cancer
Acronym: NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGS1012-C1072
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — mapatumumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Paclitaxel and carboplatin
  Interventions: Drug: Paclitaxel; Drug: Carboplatin
- B (Experimental): Paclitaxel, carboplatin and Mapatumumab 10 mg/kg
  Interventions: Biological: Mapatumumab; Drug: Paclitaxel; Drug: Carboplatin
- C (Experimental): Paclitaxel, carboplatin and Mapatumumab 30 mg/kg
  Interventions: Biological: Mapatumumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Biological: Mapatumumab — 30 mg/kg IV (in the vein), on day 1 of each 21 day cycle
  Arms: C
Biological: Mapatumumab — 10 mg/kg IV (in the vein), on day 1 of each 21 day cycle
  Arms: B
Drug: Paclitaxel — 200 mg/m^2 IV (in the vein), on day 1 of each 21 day cycle
  Other Names: Tax01; Paxene
Drug: Carboplatin — AUC 6.0 mg min/ml IV (in the vein), on day 1 of each 21 day cycle
  Other Names: Paraplatin

SUMMARY:
The purpose of this study is to evaluate the efficacy (disease response) and safety of mapatumumab in combination with carboplatin and paclitaxel as first line therapy in subjects with advanced non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed stage IIIB or stage IV advanced primary non-small cell lung cancinoma
* Age 18 years or older

Exclusion Criteria:

* Received investigational (not yet approved by a regulatory authority) or non-investigational agent to treat Lung Cancer
* Received radiation therapy within 4 weeks before randomization
* Major surgery within 4 weeks before randomization
* Minor surgery within 2 weeks before randomizaiton
* Systemic steroids within 1 week before randomization
* Any grade 2 or greater neuropathy
* History of severe (Grade 4) hypersensitivity reaction to products containing Cremophor EL (cyclosporine, teniposide)
* History of any infection requiring hospitalization or antibiotics within 2 weeks before randomization
* Known brain or spinal cord metastases
* History of other cancers within 5 years before randomization
* Known HIV, hepatitis-B or hepatitis-C infection
* Pregnant or breast-feeding women
* Previously treated with Mapatumumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2007-01; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Objective response and Progression free survival | 6 cycles, or until disease progression or unacceptable toxicity develops

SECONDARY OUTCOMES:
Disease control; Overall survival; Response duration and time to response in responders; Frequency and severity of treatment-emergent adverse events; Laboratory parameters; and Serum mapatumumab concentrations for use in a PK analysis. | 6 cycles, or until disease progression or unacceptable toxicity develops

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (33):
- United States (16):
  - Birmingham Hematology and Oncology Associates, LLC, Birmingham, Alabama
  - Desert Hematology Oncology Medical Group, Inc., Rancho Mirage, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Osceola Cancer Center, Kissimmee, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Rush University Medical Center, Chicago, Illinois
  - LaGrange Oncology Associates, LaGrange, Illinois
  - Orchard Research, LLC, Skokie, Illinois
  - Kentuckiana Cancer Institute, PLLC, Louisville, Kentucky
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - Chevy Chase Health Care, Chevy Chase, Maryland
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Medical University of South Carolina: Hollings Cancer Center, Charleston, South Carolina
  - The Sarah Cannon Cancer Center, Nashville, Tennessee
  - UT Health Science Center at San Antonio, Be Well Center, San Antonio, Texas
  - Fairfax-Northern Virginia Hematology Oncology, PC, Fairfax, Virginia
- Germany (10):
  - Charite - Campus Mitte, Universitätsmedizin Berlin, Abteilung Onkologie und Hämatologie, Berlin
  - Universitätsmedizin Berlin, Centrum für Innere Medizin, Berlin
  - Asklepios Fachkliniken München-Gauting, Gauting
  - Krankenhaus Großhansdorf, Großhansdorf
  - Krankenhaus Martha-Maria Halle-Dölau, Halle
  - Universitätsklinik Magdeburg, Klinik für Kardiologie, Angiologie und Pneumologie, Magdeburg
  - Klinikum der Johannes-Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Mannheim, Chirurgische Klinik, Mannheim
  - Pius-Hospital, Oldenburg
  - Paracelsus Klinik, Zentrum für Tumordiagnostik und -therapie, Osnabrück
- Hungary (4):
  - Fővárosi Önkormányzat Uzsoki Utcai Kórház, Budapest
  - Országos Korányi TBC és Pulmonológiai Intezet, Budapest
  - Debrecen University, Medical and Health Center, Dept of Oncology, Debrecen
  - Kenézy Gyula Kórház, Debrecen, Pulmonológia, Debrecen
- Romania (3):
  - Institutul Oncologic 'Prof Dr. Al Trestioreanu' Bucuresti, Bucharest
  - Institutul Oncologic 'Prof . Dr. I. Chiricuta' Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic Judetean Oradea, Oncology Department, Oradea

REFERENCES:
- [Derived] von Pawel J, Harvey JH, Spigel DR, Dediu M, Reck M, Cebotaru CL, Humphreys RC, Gribbin MJ, Fox NL, Camidge DR. Phase II trial of mapatumumab, a fully human agonist monoclonal antibody to tumor necrosis factor-related apoptosis-inducing ligand receptor 1 (TRAIL-R1), in combination with paclitaxel and carboplatin in patients with advanced non-small-cell lung cancer. Clin Lung Cancer. 2014 May;15(3):188-196.e2. doi: 10.1016/j.cllc.2013.12.005. Epub 2013 Dec 27. PMID 24560012